CLINICAL TRIAL: NCT01541852
Title: An Evaluation Of Losmapimod in Patients With Chronic Obstructive Pulmonary Disease (COPD) With Systemic Inflammation Stratified Using Fibrinogen (EVOLUTION)
Brief Title: Losmapimod in Chronic Obstructive Pulmonary Disease Patients Stratified by Fibrinogen.
Acronym: EVOLUTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Technology Strategy Board, United Kingdom (Other); GlaxoSmithKline (Industry); Royal Brompton & Harefield NHS Foundation Trust (Other); University of Cambridge (Other)
Responsible Party: Principal Investigator, Dr Ian B Wilkinson, Reader & Hon. Consultant Physician, Clinical Pharmacology/GIM, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A092519; 2011-004936-75 (EudraCT Number)
Record Dates: First submitted 2012-02-20; First posted 2012-03-01 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Vascular Inflammation; FDG PET-CT; COPD; Atherosclerosis; p38 MAP kinase inhibitor
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Atherosclerosis | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Losmapimod (Active Comparator): 7.5mg tablet twice daily
  Interventions: Drug: Losmapimod
- Placebo (Placebo Comparator): One tablet twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losmapimod — One tablet of Losmapimod 7.5mg twice daily
  Other Names: GW856553
  Arms: Losmapimod
Drug: Placebo — One tablet twice daily
  Other Names: Lactose Monohydrate
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine the effect of Losmapimod on blood vessels in patients with Chronic Obstructive Pulmonary Disease (COPD). Although COPD is a lung disease, it is also associated with an increased risk of cardiovascular disease (e.g. heart attacks and stroke). The investigators believe that this is a result of inflammation within the body, which damages the lining (endothelium) and walls of blood vessels. These changes can promote the development of fatty deposits within the walls of arteries (atherosclerosis) which can rupture and block arteries causing damage.

DETAILED DESCRIPTION:
The study aims to enrol sufficient COPD subjects (stratified by fibrinogen level) so that 60 patients complete the study. Study patients will have a 50% chance of receiving either Losmapimod or Placebo. Patients will be expected to attend for up to 12 visits, over a 24 week period. The visits consist of an initial screening visit, and 2 pre-dose imaging visits to include a PET-CT scan and an optional MRI scan. The next 7 visits (at 2-4 weekly intervals) involve blood tests and safety evaluations. A number of procedures including heart tracings (ECGs), non-invasive vascular measurements and lung function tests at the start and at the end of the study. Repeat imaging with PET-CT and MRI will be performed at the end of the study and a follow-up visit.

The purpose of the study is to see if the study medication has a beneficial effect on vascular function and structure. It is envisaged that this trial will help define more evolutionary biomarkers to focus on to help COPD patients in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 50 and 85 years of age inclusive at screening, with a body weight ≥ 45 kg and BMI ≤35 kg/m2.
2. Patients with a clinical diagnosis of COPD with GOLD Stages 1, 2, 3 or 4, or GOLD-U.
3. Patient has FEV1/FVC < 0.7 post-bronchodilator.
4. Patient is a smoker or an ex-smoker with a smoking history of at least 10 pack years (1 pack year = 20 cigarettes smoked per day for 1 year or equivalent).
5. Baseline fibrinogen value of >2.8 g/L (Klauss method)
6. ALT < 2xULN at screening; alkaline phosphatase and bilirubin > 1.5xULN at screening (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
7. Patients must have a QTc <450 msec on screening (V1) ECG (using average value of triplicate ECGs). For patients with complete Right bundle branch block, the QTc must be <480msec on Screening V1 ECG. Patients with other ECG findings will be excluded if warranted at the discretion of the CI/PI. QTc readings will be QTcF.
8. Patients who fulfil local imaging centre requirements will be enrolled.

Exclusion Criteria:

The presence of any of the following will preclude patient inclusion:

1. Inability in the opinion of the PI to provide Informed Consent.
2. A cardiovascular event in the last 6 months (i.e. acute coronary syndrome, unstable angina, CABG, PCI, stroke, MI, carotid endarterectomy).
3. Patients on daunorubicin, doxorubicin, topotecan, mitoxantrone.
4. Previous lung reduction surgery.
5. Patients with known clinically significant pulmonary diagnoses in which inflammation is thought to play a role including diagnosis of bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung disease, or α1-antitrypsin deficiency.
6. A positive pre-trial Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
7. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
8. Patients with known chronic infections such as HIV or known active tuberculosis.
9. Patients with rheumatoid arthritis, connective tissue disorders and other conditions known to be associated with active chronic inflammation (e.g. Inflammatory Bowel Disease).
10. Insulin controlled Type 1 or Type 2 diabetics.
11. Diabetics on oral hypoglycaemics/diet with HbA1c (DCCT) > 8% (OR HbA1c (IFCC) > 64 mmol/mol), at screening. [note: fasting glucose to be checked again at first FDG-PET/CT scan, and if glucose > 11mmol/L at that visit, patients will be excluded from trial]
12. Participation in a previous research trial in the last 3 years which involved exposure to significant ionising radiation (i.e. cumulative research radiation dose >5 mSv)
13. History of malignancy within the past 5 years (with the exception of localized carcinoma of the skin that has been resected for cure).
14. Previous exposure to Losmapimod.
15. Patients who have donated more than 500 mL of blood within 2 months prior to the trial medication administration, Visit 3 (Day 1).
16. Participation in a clinical trial where the patient has received a drug or new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of the drug (whichever is longer) prior to the first dose of trial medication, Visit 3 (Day 1).
17. History of alcohol/drug abuse or dependence within 6 months of the trial, Screening Visit 1 (Day -45 to -14).
18. Women of childbearing potential are excluded from this trial.
19. Any medical history or clinically relevant abnormality that is deemed by the principal investigator and/or medical monitor to make the patient ineligible for inclusion because of a safety concern.
20. Use of systemic corticosteroids (oral or IV) 4 weeks prior to Visit 2 (Day -14 to -1).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Vascular inflammation on FDG PET-CT | Days 0 to Day 112
  To determine the effect of Losmapimod in COPD patients on vascular structure and function as assessed by the change in Vascular inflammation as measured by FDG PET-CT
Endothelial function as measured by flow mediated dilatation | Days 0 to Day 112
  To determine the effect of Losmapimod in COPD patients on vascular structure and function as assessed by the change in endothelial function as measured by flow mediated dilatation
Arterial structure and plaque characteristics on MRI | Days 0 to Day 112
  To determine the effect of Losmapimod in COPD patients on vascular structure and function as assessed by the change in arterial structure and plaque characteristics as measured by MRI (MRI is an optional sub-study and analysis will be based on a sufficient number of datasets).

SECONDARY OUTCOMES:
Lung inflammation on FDG PET-CT | Days 0 to 112
  To determine the effects of Losmapimod on the change in inflammation in lung tissue as assessed by FDG PET-CT
Fat inflammation on FDG PET-CT | Days 0 to 112
  To determine the effects of Losmapimod on the change in fat inflammation as assessed by FDG PET-CT
Arterial stiffness as measured by arterial tonometry | Days 0 to 112
  To determine the effects of Losmapimod on the change in arterial stiffness as measured by arterial tonometry
Blood biomarkers of systemic inflammation (Fibrinogen and high sensitivity CRP) | Days 0 to 112
  To determine the effects of Losmapimod on the change in blood biomarkers of inflammation such as Fibrinogen and high sensitivity CRP
Indices of lung function (6 minute walk test and sniff nasal inspiratory pressure) | Days 0 to 112
  To determine the effects of Losmapimod on the change in indices of lung function and physical performance as measured by 6 minute walk test and sniff nasal inspiratory pressure
Body composition and fat as assessed by Free fat mass index | Days 0 to 112
  To determine the effects of Losmapimod on the change in body composition and fat as measured by Free fat mass index
Number of adverse events as a measure of safety and tolerability | Days 0 to 112
  To determine the effects of Losmapimod on the number of adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cheriyan, MD, Principal Investigator — Cambridge University Hospitals; Michael Polkey, MD, Principal Investigator — Royal Brompton & Harefield Foundation NHS Trust
Locations (2):
- United Kingdom (2):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - Royal Brompton & Harefield NHS Foundation Trust, London, London